CLINICAL TRIAL: NCT02169206
Title: Clinical Trial on Frozen Shoulder Using Bilateral Shoulder Radiography in Different Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir Reza Kachooei, M.D., Mashhad University of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 910177
Record Dates: First submitted 2014-06-19; First posted 2014-06-23 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Frozen Shoulder
Keywords: Frozen shoulder; scapulothoracic angle; scapulohumeral angle; acromiohumeral distance; center equator distance; shoulder radiography
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- shoulder radiography (Other): Bilateral shoulder AP standard plain x-ray in 0 and 90 degrees of arm abduction. Non-affected shoulder is used to be compared with the affected shoulder.
  Interventions: Radiation: Bilateral shoulder anteroposterior radiography

INTERVENTIONS:
Radiation: Bilateral shoulder anteroposterior radiography — 1. Patient standing with the tube in front and 105 cm far from the shoulder radiating perpendicular to the cassette in the back, both arms hanging aside the trunk in 0 degrees of arm abduction, 0 degrees of rotation and 0 degrees of extension with the thumb facing forward to obtain true bilateral shoulder anteroposterior view. Voltage and exposure time differs regarding each person's body mass.
  2. In the same position, the patient only elevates the arm up to 90 degrees of abduction.

SUMMARY:
This study on frozen shoulder addressed the null hypothesis that there is no difference in the motion of scapula against the thoracic wall between affected and non-affected shoulder.

DETAILED DESCRIPTION:
Adult patients with unilateral shoulder pain lasted for more than one month, accompanied by passive and active limitation of range of motion in all directions will be included. Patients with bilateral involvement, history of trauma, history of surgery on the affected shoulder, history of fracture, shoulder osteoarthritis, symptoms less than one month and any signs of rotator cuff tear will be excluded. MR imaging will be done to exclude other pathologies and frank rotator cuff tear.

ELIGIBILITY:
Inclusion Criteria:

* adult patients with unilateral shoulder pain lasted for more than one month, accompanied by passive and active limitation of range of motion in all directions

Exclusion Criteria:

* bilateral involvement, history of trauma, history of surgery on the affected shoulder, history of fracture, shoulder osteoarthritis, symptoms less than one month and any signs of rotator cuff tear. MRI will be done to rull out the rotator cuff tear.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-10; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Radiographic parameter (scapulothoracic angle) measured in angle | one year

OTHER OUTCOMES:
Center equator distance | one year
  Center-equator distance (CED): On radiography, the humeral head center (HHC) is determined using a circular template. A perpendicular line to glenoid is drawn passing through its middle point which supposed to be the glenoid equator line (GEL). The distance between the HHC and GEL is measured in millimeters and considered positive if HHC is above and negative if HHC is below the GEL.
Scapulohumeral angle | one year
  Scapulohumeral angle (SHA): The angle formed between humeral shaft axis and lateral border of scapula starting from the inferior angle is called scapulohumeral angle.
Acromiohumeral distance | one year
  Acromiohumeral distance (AHD): Distance between the line drawn along the acromial lower border density and the highest point of the humeral head is measured in millimeters as acromiohumeral distance (AHD).

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad H Ebrahimzadeh, M.D., Study Director — Mashhad University of Medical Sciences; Amir R Kachooei, M.D., Principal Investigator — Mashhad University of Medical Sciences
Locations (1):
- Mashhad University of Medical Sciences, Mashhad, Khorasan-Razavi, Iran